CLINICAL TRIAL: NCT05636007
Title: Early Detection of noctUrnal hypoglyCemiA in TypE 2 Diabetes Using Pulse Rate Variability Measured by a Smartwatch(EDUCATED-Smartwatch)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xiao-dong Zhuang, professor, Sun Yat-sen University
Other Study IDs: EDUCATED-Smartwatch Study
Record Dates: First submitted 2022-11-22; First posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Hypodlycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Huawei Watch — pulse rate variability measured by a smartwatch

SUMMARY:
In patients with type 2 diabetes, it is necessary to identify and manage nocturnal hypoglycemia as early as possible, so as to reduce the damage caused by nocturnal hypoglycemia.We explore whether smartwatches can provide early warning of nocturnal hypoglycemic events in patients with type 2 diabetes by detecting changes in pulse variability.

ELIGIBILITY:
Inclusion Criteria:

* 1. ≥18 years old 2.continuous glucose monitoring in patients with type 2 diabetes 3.Agreed to research into the group, and be able to sign the informed consent

Exclusion Criteria:

* 1.Arrhythmia, such as sinus arrest, sick sinus syndrome, atrial fibrillation, atrial flutter 2.Such as acute or chronic infectious diseases,hyperthyroidism and thyroid function did not return to normal pregnancy 3.nursing mothers

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: type 2 diabetes patients with continuous glucose monitoring
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
nocturnal hypoglycemia | 8 months
  hypoglycemia occuring during 0AM to 6AM

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No